CLINICAL TRIAL: NCT01248611
Title: Nasal Fentanyl for Patient Controlled Treatment of Pain in Cancer An Open Label Prospective Phase I b Study
Brief Title: Nasal Fentanyl for Patient Controlled Treatment of Pain in Cancer
Acronym: NFCP1-2010
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFCP1-2010
Record Dates: First submitted 2010-11-18; First posted 2010-11-25 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Pain; Cancer
Keywords: pain; adverse effects; safety; feasibility
MeSH Terms: conditions — Chronic Pain; Neoplasms; Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fentanyl (Experimental): cancer patients with pain
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — nasally, dose titrated to effect
  Other Names: Instanyl (nNcomed Pharma)

SUMMARY:
Traditionally cancer pain is treated with long acting opioids such as morphine around the clock. However, there is no evidence that all patients have a stable pain requiring around the clock medication. So far opioids for self-administration with a rapid onset of action have not been available. Recently a nasal formulation of fentanyl (an opioid similar to morphine) was released in Europe for treatment of breakthrough pain, i.e. an unpredictable pain with short duration that breaks through the otherwise stable pain controlled with the around the clock medication. The basic idea is that this formulation may open for patient controlled analgesia of chronic cancer pain, due to the ultra rapid onset of action of nasally delivered fentanyl. This means that the patient only takes medication when in pain. This single center feasibility / safety study is the first part of a study to investigate this alternative cancer pain treatment approach.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients with metastatic disease
2. Adult (older than 18 years)
3. Life expectancy of > 3 months
4. Cancer-related pain > 3 on an 11 point Numerical Rating Scale (NRS)
5. In the need of opioids (step II or III)
6. Able to use nasal drugs.
7. Women of child bearing potential using adequate contraception
8. Informed consent given according to applicable requirements before any trial-related activities. Trial-related activities are any procedure that would not have been performed during the routine management of the patient

Exclusion Criteria:

1. History of substance abuse
2. Cognitive impairment which makes the patient unable to complete questionnaires or not able to comply with the study procedures
3. Treated with MAO inhibitor within the last 14 days
4. Known hypersensitivity to study drug or specific contraindications to the study drug
5. Nasopharyngeal device such as gastric tube
6. Concomitant participation in any other trials dealing with pain with an investigational drug or device apart from cancer treatment within 14 days prior to inclusion in this trial
7. Pathological conditions of the nasal cavity as contraindication to nasal fentanyl
8. Sleep apnoea syndrome
9. Pregnant or breastfeeding women
10. Psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
sedation/drowsiness | 10 days
  scores on a 0-10 numerical rating scale; 0=none / 10=intolerable
nausea and vomiting | 10 days
  nausea scores on a 0-10 numerical rating scale; 0=none / 10=intolerable vomiting yes/no

SECONDARY OUTCOMES:
pain intensity | 10 days
  scores on a 0-10 numerical rating scale; 0=none / 10=intolerable

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD. PhD, Principal Investigator — St.Olav's Hospital
Locations (1):
- St.Olavs University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Thronaes M, Kaasa S, Dale O. A pilot study of nasal fentanyl for patient controlled treatment of cancer pain. J Opioid Manag. 2014 Jan-Feb;10(1):21-8. doi: 10.5055/jom.2014.0188. PMID 24604566